CLINICAL TRIAL: NCT00461097
Title: Oral Desensitization to Egg With Subsequent Induction of Tolerance for Egg-Allergic Children (CoFAR 3)
Brief Title: Oral Immunotherapy for Childhood Egg Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT CoFAR3; COFAR; U19AI066738 (NIH)
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Hypersensitivity; Immediate Hypersensitivity; Food Hypersensitivity
Keywords: Egg Allergy; Egg Oral Immunotherapy (OIT); Food Allergy
MeSH Terms: conditions — Hypersensitivity; Hypersensitivity, Immediate; Food Hypersensitivity; Egg Hypersensitivity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Egg Oral Immunotherapy (OIT) (Experimental): Subjects ingest egg white solid (EWS) on Visit 1 (initial day dose escalation up to 50 mg), followed by a build-up phase (escalating daily egg doses every 2 wks, achieving a maintenance dose by 32-40 wks). Thereafter, subjects are on a maximally tolerated daily egg dose (306 mg to 2 gm) for ≥8 wks. After wk 44, subjects are given a 5 gm Oral Food Challenge (OFC) using EWS to identify desensitized [1] subjects. Subjects/study staff are unblinded following this OFC and either continue on their egg OIT maintenance dose of 2 gm/day or are allowed to attempt escalation up to 2 gm/day for the remainder of the study (1-3 years). A 10 gm OFC to identify desensitized [1] subjects occurs at specified intervals under prescribed conditions (yrs 2 - 4). Subjects who pass this 1st 10 gm OFC stop study therapy for 4-6 wks, then have a 2nd 10 gm OFC. Subjects that pass this 2nd 10 gm OFC are considered tolerant [2], stop EWS dosing and add egg to their diet.
  Interventions: Drug: Egg oral immunotherapy
- Control Group (Placebo Comparator): Subjects ingest placebo (cornstarch) during Visit 1 (initial day of dose escalation up to 50 mg), followed by a build-up phase (escalating daily placebo doses every 2 wks, achieving a maintenance dose by 32-40 wks). Thereafter, subjects were on a maximally tolerated daily placebo dose (306 mg to 2 gm) for ≥8 wks. After wk 44, subjects were given a 5 gm Oral Food Challenge (OFC) using egg white solid to identify desensitized [1] subjects. Subjects/study staff were unblinded following this initial 5 gm OFC. After unblinding, subjects discontinued further placebo dosing and continued on an egg-restricted diet. A 10 gm OFC was administered under prescribed conditions to subjects if their egg-specific serum IgE level was below 2 kUA/L. They were followed in the study up to 2 years. [1] Desensitized: Subject does not react to egg during OFC while taking daily doses of therapy. [2] Tolerant: Subject does not react to egg during OFC 4-6 wks after abstinence from egg consumption.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Egg oral immunotherapy — Egg white solid powder
  Arms: Egg Oral Immunotherapy (OIT)
Drug: Control Group — Placebo for egg white solid
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if oral immunotherapy (OIT) will desensitize a child with an allergy to egg and eventually lead to the development of tolerance to egg.

DETAILED DESCRIPTION:
In the United States, as many as 6% to 8% of children are affected by food allergy. In young children, allergic reactions to egg can range from mild rash to systemic anaphylaxis. The usual standard of care for allergy is complete avoidance of this food allergen and treatment of accidental systemic reactions by access to self-injected epinephrine. However, accidental exposure to allergens in processed foods may be difficult to avoid. Currently, several therapeutic strategies are being investigated to prevent and treat food allergies. Since standard injection (under the skin) immunotherapy for food allergy is associated with a high rate of allergic reactions, a few studies have recently tried oral immunotherapy (OIT) in food allergy. The purpose of this study is to determine the safety and efficacy of the administration of OIT. The intent is to develop desensitization and eventually tolerance to egg allergen. This study will evaluate tolerance to egg white solid that may be gained by gradually increasing the amounts of egg white solid given to a child over a long period of time.

This study will last up to 48 months. The participants will be randomly assigned to receive oral immunotherapy treatment with egg white solid or placebo. This study will include dose escalation and maintenance followed by oral food challenge (OFC).

For participants receiving egg OIT, visit 1 consists of multiple small incremental doses of egg white solid. This is followed by 32-40 weeks of gradual dose escalation to a stable maintenance dose of egg white solid for at least 8 weeks. At approximately Week 44, participants are given an OFC using 5 grams of egg white solid to identify desensitized individuals. Participants and study staff are unblinded following this initial OFC. Maintenance egg OIT therapy is continued for an additional 1-3 years. Oral Food Challenges with 10 grams of egg white solid will be performed for participants on maintenance egg OIT at subsequent time points (approximately Week 96 and annually thereafter) to test for desensitization. If passed, a repeat OFC after being off therapy for 4-6 weeks will be performed to test for tolerance. An OFC to test for tolerance will use 10 grams of egg white solid and be followed by an open feeding of egg.

Participants receiving placebo during dose escalation and maintenance are given an OFC using 5 grams of egg white solid to test for desensitization at approximately 44 weeks. They are unblinded at that time, continue on an egg-restricted diet, and are followed until up to 2 years. These participants will only receive an OFC at a subsequent time point if their egg Immunoglobulin E (IgE) declines to be less than 2 kilounits of antibody per liter; this OFC will use 10 grams of egg white solid and be followed by an open feeding of egg.

At selected visits, blood and urine collection, physical examination, prick skin tests, and atopic dermatitis and asthma evaluations will occur.

ELIGIBILITY:
Inclusion Criteria:

* Convincing clinical history of egg allergy
* Age 6 to 18 years, with a serum IgE [UniCAP] to egg > 5 kUA/L OR
* Age 5 to 6 years, with a serum IgE [UniCAP] to egg ≥ 12kUA/L
* Parent/guardian willing to provide informed consent
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* History of severe anaphylaxis to egg. More information on this criterion can be found in the protocol.
* Known allergy to corn
* Chronic disease requiring therapy (e.g., heart disease, diabetes). Participants who have asthma, atopic dermatitis, or rhinitis are not excluded.
* Participation in any interventional study for the treatment of food allergy in the 6 months prior to study entry
* Participant is on "build-up phase" of immunotherapy and has not reached maintenance dosing. Participants tolerating maintenance allergen immunotherapy are not excluded.
* Severe asthma, uncontrolled mild or moderate asthma. More information on this criterion can be found in the protocol.
* Inability to discontinue antihistamines for the initial day of escalation, skin testing, and OFC
* Omalizumab or other nontraditional forms of oral or sublingual allergen immunotherapy, immunomodulator therapy, or biologic therapy in the 12 months prior to study entry. Participants who have taken corticosteroids are not excluded.
* Investigational drugs 90 days prior to study entry or planned use of an investigational drug during the study period
* Pregnancy or breastfeeding

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Study Chair — University of North Carolina; Stacie Jones, MD, Study Chair — Allergy/Immunology Department, Arkansas Children's Hospital; Robert Wood, MD, Principal Investigator — Johns Hopkins University; Scott Sicherer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; David Fleischer, MD, Principal Investigator — National Jewish Health
Locations (5):
- United States (5):
  - University of Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - National Jewish Medical and Research Center, Denver, Colorado
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hills, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Baral VR, Hourihane JO. Food allergy in children. Postgrad Med J. 2005 Nov;81(961):693-701. doi: 10.1136/pgmj.2004.030288. PMID 16272231
- [Background] Sicherer SH, Sampson HA. 9. Food allergy. J Allergy Clin Immunol. 2006 Feb;117(2 Suppl Mini-Primer):S470-5. doi: 10.1016/j.jaci.2005.05.048. PMID 16455349
- [Background] Wood RA. The natural history of food allergy. Pediatrics. 2003 Jun;111(6 Pt 3):1631-7. PMID 12777603
- [Result] Burks AW, Jones SM, Wood RA, Fleischer DM, Sicherer SH, Lindblad RW, Stablein D, Henning AK, Vickery BP, Liu AH, Scurlock AM, Shreffler WG, Plaut M, Sampson HA; Consortium of Food Allergy Research (CoFAR). Oral immunotherapy for treatment of egg allergy in children. N Engl J Med. 2012 Jul 19;367(3):233-43. doi: 10.1056/NEJMoa1200435. PMID 22808958
- [Derived] Jones SM, Burks AW, Keet C, Vickery BP, Scurlock AM, Wood RA, Liu AH, Sicherer SH, Henning AK, Lindblad RW, Dawson P, Berin C, Fleischer DM, Leung DYM, Plaut M, Sampson HA; Consortium of Food Allergy Research (CoFAR). Long-term treatment with egg oral immunotherapy enhances sustained unresponsiveness that persists after cessation of therapy. J Allergy Clin Immunol. 2016 Apr;137(4):1117-1127.e10. doi: 10.1016/j.jaci.2015.12.1316. Epub 2016 Mar 9. PMID 26924470
- Available data/document: Individual Participant Data Set: SDY218 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY218 — ImmPort study identifier is SDY218
- Available data/document: Study summary, -design, -adverse events, -demographics,-lab tests,-mechanistic assays, -study files: SDY218 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY218 — ImmPort study identifier is SDY218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at five university-based medical centers in the United States (Mt. Sinai School of Medicine, Johns Hopkins University, Duke University, National Jewish Medical Center, University of Arkansas Children's Hospital) from July 2007 to December 2008.
Groups:
- Placebo: Subjects ingest placebo (cornstarch) during Visit 1 (initial day of dose escalation up to 50 mg), followed by a build-up phase (escalating daily placebo doses every 2 wks, achieving a maintenance dose by 32-40 wks). Thereafter, subjects were on a maximally tolerated daily placebo dose (306 mg to 2 gm) for ≥8 wks. After wk 44, subjects were given a 5 gm Oral Food Challenge (OFC) using egg white solid to identify desensitized [1] subjects. Subjects/study staff were unblinded following this initial 5 gm OFC. After unblinding, subjects discontinued further placebo dosing and continued on an egg-restricted diet. A 10 gm OFC was administered under prescribed conditions to subjects if their egg-specific serum IgE level was below 2 kUA/L. They were followed in the study up to 2 years. [1] Desensitized: Subject does not react to egg during OFC while taking daily doses of therapy. [2] Tolerant: Subject does not react to egg during OFC 4-6 wks after abstinence from egg consumption.
Period: Overall Study
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Started | 40 | 15
Had Month 10 (Wk 44) Oral Food Challenge | 35 | 13
Had Month 22 (Wk 96) Oral Food Challenge | 34 | 1
Had Year 3 (Mnth 36) Oral Food Challenge | 16 | 0
Had Year 4 (Mnth 48) Oral Food Challenge | 7 | 0
Completed | 40 (Completed: Participants who were assessed for the primary outcome measure and outcome measure #6.) | 15 (Completed: Participants who were assessed for the primary outcome measure.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo | Total
Number analyzed (Participants) | 40 | 15 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 15 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.1 (1.6) | 7.1 (1.6) | 7.1 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 25 | 9 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 38 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 34 | 14 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 15 | 55
Atopic Dermatitis Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Atopic Dermatitis Total Score is scored on a 10 point scale from 0 to 9 where a higher score indicates increased severity of atopic dermatitis. This score is a combination of 3 scores that range from 0 to 3 in the following areas: body surface area score, disease course, and disease intensity.
  Scores on a scale | 3.1 (2.5) | 3.0 (2.8) | 3.1 (2.5)
Total IgE [Mean (Standard Deviation); unit: kU/L] — Total amount of serum immunoglobulin E. Individuals who are not allergic may have a total IgE as high as 304 kU/L.
  kU/L | 1378.7 (1728.6) | 1464.7 (1182.7) | 1402.1 (1588.1)
Egg IgE [Mean (Standard Deviation); unit: kUA/L] — Amount of serum egg-specific immunoglobulin E. Individuals with an egg IgE of <0.35 kUA/L are considered not to be sensitized to egg.
  kUA/L | 32.9 (54.7) | 32.1 (27.3) | 32.7 (48.5)
Egg Skin Prick Test Score [Mean (Standard Deviation); unit: mm] — This score is calculated by subtracting the size of the saline wheal (in mm) from the size of the egg wheal (in mm) observed for a skin prick test. Individuals with an egg skin prick test score of < 3 mm are considered to have a negative result.
  mm | 11.8 (5.7) | 12.8 (4.3) | 12.1 (5.4)
Age at Initial Egg Allergic Reaction [Mean (Standard Deviation); unit: years] | 2.3 (2.1) | 1.3 (1.4) | 2.0 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Successfully Consumed 10,000 mg of Egg White Solid Followed by Open Feeding of Egg
Description: Tolerance Assessment: Participants who successfully consumed without dose-limiting symptoms 10,000 mg of egg white solid during a double-blind placebo-controlled oral food challenge were then given an open feeding of egg and those who successfully consumed the open feeding of egg were counted as successes.
Time Frame: At the 2 year time point; Egg OIT participants must be approximately 4-6 weeks post-discontinuation of therapy
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Number analyzed (Participants) | 40 | 15
percentage of participants | 27.5 | 0
Statistical Analysis 1: Comparison: Egg Oral Immunotherapy (OIT) vs Placebo; Number of participants who successfully consumed 10,000 mg of egg white solid was compared using Barnard's statistic with the null hypothesis that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.025, Barnard's statistic — No adjustments were made to the p-value; The a priori threshold for statistical significance is 0.05; Risk Difference (RD) = 27.5, 95% CI 2-sided [4.3 to 43.9]

2. Secondary Outcome: Percent of Participants Who Successfully Consumed 5,000 mg of Egg White Solid
Description: Desensitization assessment: Participants who successfully consumed without dose-limiting symptoms 5,000 mg of egg white solid during a double-blind placebo-controlled oral food challenge were counted as successes.
Time Frame: Following the blinded desensitization phase at approximately Week 44
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Number analyzed (Participants) | 40 | 15
percentage of participants | 55.0 | 0.0

3. Secondary Outcome: Percent of Participants Who Successfully Consumed a 50 mg Dose at Initial Escalation
Description: On the initial day of dosing, participants were offered 0.1 mg of egg white solid or placebo followed by an approximate doubling every 30 minutes up to a 50 mg dose providing limiting reactions do not occur.
Time Frame: Initial day of dosing
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Number analyzed (Participants) | 40 | 15
percentage of participants | 22.5 | 86.7

4. Secondary Outcome: Percent of Participants Who Achieved a Maintenance Dose of 2,000 mg
Description: For participants whose maximum tolerated dose on the initial escalation day was less than 50 mg, doses were doubled every 2 weeks up to 50 mg. After 50 mg, dosing was increased to 75 mg, and then dosing increased by 25% until the 2000 mg dose was reached. The maximum time allowed for the build-up phase was 40 weeks; the dose achieved at 40 weeks was considered the maintenance dose.
Time Frame: Following the blinded desensitization phase at approximately Week 44
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Number analyzed (Participants) | 40 | 15
percentage of participants | 45.0 | 80.0

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: This study graded the severity of Adverse Events experienced by participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.
Time Frame: Baseline through the 2-year primary endpoint
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: participants
Arm/Group | Egg Oral Immunotherapy (OIT) | Placebo
Number analyzed (Participants) | 40 | 15
participants | 3 | 0

6. Secondary Outcome: Percent of Participants in the Egg OIT Treatment Arm Who Successfully Consumed 10,000 mg of Egg White Solid
Description: Tolerance Assessment: Participants in the Egg OIT treatment arm who were not tolerant at 2 years were offered an additional 2 years of therapy. A 10,000 mg double-blind placebo controlled oral food challenge to egg was done the same way as the one performed at 2 years for these participants in order to identify tolerant individuals in the 2 to 4 year extension segment. The tolerant individuals from this segment were then added to the tolerant individuals from the 2 year segment.
Time Frame: 4 years (48 months)
Measure: Number; unit: percentage of participants
Arm/Group | Egg Oral Immunotherapy (OIT)
Number analyzed (Participants) | 40
percentage of participants | 52.5

ADVERSE EVENTS:
Time Frame: Baseline through 2 year primary endpoint for Egg OIT and Placebo groups; then for Egg OIT only from 2 to 4 years.
Description: This study graded the severity of Adverse Events experienced by participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.
Groups:
- Egg Oral Immunotherapy (OIT), 0-2 Years: Subjects ingest egg white solid (EWS) on Visit 1 (initial day dose escalation up to 50 mg), followed by a build-up phase (escalating daily egg doses every 2 wks, achieving a maintenance dose by 32-40 wks). Thereafter, subjects are on a maximally tolerated daily egg dose (306 mg to 2 gm) for ≥8 wks. After wk 44, subjects are given a 5 gm Oral Food Challenge (OFC) using EWS to identify desensitized [1] subjects. Subjects/study staff are unblinded following this OFC and either continue on their egg OIT maintenance dose of 2 gm/day or are allowed to attempt escalation up to 2 gm/day. A 10 gm OFC to identify desensitized [1] subjects occurs at month 22. Subjects who pass this 1st 10 gm OFC stop study therapy for 4-6 wks, then have a 2nd 10 gm OFC at year 2. Subjects that pass this 2nd 10 gm OFC are considered tolerant [2], stop EWS dosing and add egg to their diet.
- Placebo, 0-2 Years: Subjects ingest placebo (cornstarch) during Visit 1 (initial day of dose escalation up to 50 mg), followed by a build-up phase (escalating daily placebo doses every 2 wks, achieving a maintenance dose by 32-40 wks). Thereafter, subjects were on a maximally tolerated daily placebo dose (306 mg to 2 gm) for ≥8 wks. After wk 44, subjects were given a 5 gm Oral Food Challenge (OFC) using egg white solid to identify desensitized [1] subjects. Subjects/study staff were unblinded following this initial 5 gm OFC. After unblinding, subjects discontinued further placebo dosing and continued on an egg-restricted diet. A 10 gm OFC was administered under prescribed conditions to subjects if their egg-specific serum IgE level was below 2 kUA/L. They were followed in the study up to 2 years. [1] Desensitized: Subject does not react to egg during OFC while taking daily doses of therapy. [2] Tolerant: Subject does not react to egg during OFC 4-6 wks after abstinence from egg consumption.
- Egg Oral Immunotherapy (OIT), 2-4 Years: Subjects who failed the 1st or 2nd 10 gm OFC at month 22 or year 2 continue on their egg OIT maintenance dose of 2 gm/day of egg white solid (EWS) or are allowed to attempt escalation up to 2 gm/day for the remainder of the study. Subjects who are not considered tolerant may have a 10 gm OFC at year 3 and year 4 to assess desensitization. Subjects who pass the 1st 10 gm OFC stop study therapy for 4-6 wks, then have a 2nd 10 gm OFC. Subjects that pass this 2nd 10 gm OFC are considered tolerant [2], stop EWS dosing and add egg to their diet.
  Note: The total number of subjects assessed for non-systematic adverse events was 36 (subjects with post 2-year follow-up) and for systematic adverse events was 22 (subjects with post 2-year dosing).
Arm/Group | Egg Oral Immunotherapy (OIT), 0-2 Years | Placebo, 0-2 Years | Egg Oral Immunotherapy (OIT), 2-4 Years
Serious Adverse Events (participants affected / at risk) | 3/40 | 0/15 | 1/36
Other Adverse Events (participants affected / at risk) | 40/40 | 15/15 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Egg Oral Immunotherapy (OIT), 0-2 Years (N=40) | Placebo, 0-2 Years (N=15) | Egg Oral Immunotherapy (OIT), 2-4 Years (N=36)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Egg Oral Immunotherapy (OIT), 0-2 Years (N=40) | Placebo, 0-2 Years (N=15) | Egg Oral Immunotherapy (OIT), 2-4 Years (N=36)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0/22 (0)
Eye pruritus (Eye disorders) | 5 (71) | 3 (4) | 1/22 (11)
Lacrimation increased (Eye disorders) | 3 (5) | 0 (0) | 0/22 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0/22 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4)
Vomiting (Gastrointestinal disorders) | 10 (15) | 2 (2) | 6 (8)
Abdominal discomfort (Gastrointestinal disorders) | 34 (807) | 4 (9) | 4/22 (20)
Abdominal pain (Gastrointestinal disorders) | 16 (28) | 2 (2) | 0/22 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (20) | 0 (0) | 1/22 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/22 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (79) | 0 (0) | 0/22 (0)
Lip swelling (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1/22 (3)
Oral disorder (Gastrointestinal disorders) | 31 (2457) | 3 (9) | 8/22 (214)
Vomiting (Gastrointestinal disorders) | 28 (125) | 2 (4) | 4/22 (4)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 4 (7) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (11) | 1 (1) | 8 (16)
Chest discomfort (General disorders) | 6 (8) | 0 (0) | 0/22 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0/22 (0)
Fatigue (General disorders) | 3 (6) | 0 (0) | 0/22 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0/22 (0)
Hypersensitivity (Immune system disorders) | 4 (7) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 12 (17) | 3 (3) | 6 (6)
Impetigo (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Influenza (Infections and infestations) | 11 (12) | 3 (4) | 4 (5)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (32) | 5 (12) | 6 (11)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 4 (6) | 4 (4) | 5 (8)
Pharyngitis streptococcal (Infections and infestations) | 4 (11) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 8 (13) | 2 (3) | 5 (7)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 20 (59) | 9 (10) | 10 (19)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (2) | 4 (4)
Headache (Nervous system disorders) | 3 (25) | 2 (2) | 1/22 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0/22 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 2 (2) | 6 (8)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 1 (1) | 4 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 1 (1) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (182) | 5 (35) | 3/22 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0/22 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0/22 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0/22 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 (385) | 5 (27) | 2/22 (151)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 2 (2) | 0/22 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 22 (658) | 1 (1) | 4/22 (36)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 21 (72) | 6 (54) | 1/22 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 0 (0) | 0/22 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 1 (1) | 0/22 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (42) | 0 (0) | 0/22 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0/22 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0/22 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (424) | 3 (12) | 4/22 (78)
Rash (Skin and subcutaneous tissue disorders) | 4 (9) | 3 (14) | 0/22 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0/22 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 27 (398) | 5 (19) | 5/22 (18)
Flushing (Vascular disorders) | 18 (43) | 3 (3) | 2/22 (2)
Ear discomfort (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 0/22 (0)
Ear pruritus (Ear and labyrinth disorders) | 3 (10) | 0 (0) | 0/22 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0/22 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0/22 (0)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (5)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0/22 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No